CLINICAL TRIAL: NCT06375460
Title: Real-time Engagement for Learning to Effectively Control Type 2 Diabetes
Acronym: REFLECT2D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Dartmouth College (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); San Diego State University (Other); Emory University (Other)
Responsible Party: Principal Investigator, Mary Ellen Vajravelu, MD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24020141; 1R01DK137803-01A1 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-04-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2; Lifestyle; Hyperglycemia; Physical Inactivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Subjects will wear a continuous glucose monitor and activity watch for study duration. Subjects will be micro-randomized once daily for 90 days to receive app prompts regarding nutrition or physical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Physical Activity Focused App Prompt (Experimental): The app prompts will ask participants what went well, or did not go well with their physical activity in the previous 24 hours in relation to their blood glucose numbers.
  Interventions: Behavioral: Focused App Prompt
- Diet Focused App Prompt (Experimental): The app prompts will ask participants what went well, or did not go well with their diet in the previous 24 hours in relation to their blood glucose numbers.
  Interventions: Behavioral: Focused App Prompt
- No App Prompt (Experimental): No app prompt will be sent to the participant
  Interventions: Behavioral: No App Prompt
- Outreach for Missing Data (Experimental): Participants will be randomized to receive proactive outreach by the study team in the case of 3 or more days of missing CGM data, versus no proactive outreach
  Interventions: Behavioral: Outreach for Missing Data

INTERVENTIONS:
Behavioral: Focused App Prompt — Prompts are designed to develop knowledge and self-efficacy in diabetes-related health behaviors (capability). The paired glycemic and behavior data will provide the opportunity to reflect and to plan diet or exercise for the following day (self-reflective motivation).
  Arms: Diet Focused App Prompt; Physical Activity Focused App Prompt
Behavioral: No App Prompt — No app prompts are designed to assess whether health behaviors are affected without being prompted to reflect and change those behaviors related to glycemic control.
  Arms: No App Prompt
Behavioral: Outreach for Missing Data — For participants randomized to proactive outreach, after 3 or more days of missing CGM data, the study team will reach out to participants by phone and/or text message to troubleshoot and support participants in re-connecting with CGM and apps. For participants randomized to not receive proactive outreach, participants will be instructed to reach out to the study team at their discretion when help is needed related to CGM or app connection.
  Arms: Outreach for Missing Data

SUMMARY:
This is a clinical trial that includes a run-in period, a 90 day micro-randomized trial, and a 90-day observational period. The goal of this study is to evaluate whether providing paired real time glycemic and health behavior data in a smartphone app leads to better glycemic control among adolescents and young adults with T2D. Glycemic control will be monitored using Continuous Glucose Monitors (CGM), and health behavior data will be collected via a Fitbit activity tracker and a research app (Healthmine). Participants will be prompted to view and reflect on glycemic trends and health behavior data (Fitbit data, logging of diet and medication adherence) during the 90-day micro-randomized trial period, then observed for ongoing use of the Healthmine app and engagement with CGM in the following 90-day observation period.

DETAILED DESCRIPTION:
The objective of REFLECT2D (Real-time Engagement For Learning to Effectively Control Type 2 Diabetes) is to evaluate whether pairing real-time glycemic and health behavior data leads to improved glycemic control among adolescents and young adults with type 2 diabetes. Participants will use a mobile app that integrates continuous glucose monitor data, Fitbit activity tracker data, and diet logging, with the aim of increasing capability to interpret glycemic data (including impacts of physical activity and dietary intake), providing opportunity to plan and implement behavior change, and increasing motivation to engage in health behaviors. After a session with a Registered Dietitian and Diabetes Educator who will support participants in forming diet and activity goals, a 90-day micro-randomized trial (MRT) period will involve once daily randomization of each participant to: 1) physical-activity focused prompt, 2) dietary intake-focused prompt, or 3) no prompt. Prompts will include reviews of glycemic trends in the past 24 hours (e.g., periods of hyperglycemia, max glucose) and will ask participants to use visual summaries of activity or diet and glucose to reflect on and revise their behavioral management goals as needed. After the MRT, a 90-day observation period without prompts but with ongoing availability of continuous glucose monitor data, Fitbit, and Healthmine app will examine persistence of glycemic and behavior changes. In addition to daily micro-randomization, participants will be randomized 1:1 at study start to proactive outreach from the study team in the case of 3 or more days of missing data, versus no outreach for missing data.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes: negative diabetes autoantibodies, no suspicion for monogenic diabetes
* HbA1c ≥7.0%, stable medication use
* HbA1c 6.0-6.9% without short-acting insulin, any other stable diabetes medication use
* English-speaking (app in English)

Exclusion Criteria:

* Current pregnancy
* Hydroxyurea use (CGM sensor inaccuracies)
* Cognitive impairment or severe psychiatric condition that could interfere with participation in behavioral intervention for diabetes self-management
* Current or previously diagnosed eating disorder

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Glucose time above 180mg/dL | daily during micro randomized trial, 90 days
  measured using continuous glucose monitor
Mean daily glucose | daily during micro randomized trial, 90 days
  measured using continuous glucose monitor; mg/dL
Maximum daily glucose | daily during micro randomized trial, 90 days
  measured using continuous glucose monitor; mg/dL
Minimum daily glucose | daily during micro randomized trial, 90 days
  measured using continuous glucose monitor; mg/dL
Glucose coefficient of variability | daily during micro randomized trial, 90 days
  measured using continuous glucose monitor
Mean amplitude of glycemic excursions | daily during micro randomized trial, 90 days
  measured using continuous glucose monitor
Hemoglobin A1c | through study completion, 6 months average
  lab-based measure to assess longer-term glycemic control, collected at study visit
Fasting glucose | through study completion, 6 months average
  lab-based measure to assess glycemic control, collected at study visit
Objective physical activity (step count) | daily during micro randomized trial, 90 days;
  step count measured using the Fitbit physical activity tracker
Objective physical activity (moderate-vigorous physical activity) | daily during micro randomized trial, 90 days;
  moderate-vigorous physical activity (>100 steps per minute) will be measured using Fitbit activity tracker
Self-reported physical activity | through study completion, 6 months average
  assessed using PACE+ Adolescent Physical Activity Measure (PACE+) questionnaire to determine days with at least 60 minutes of moderate-vigorous physical activity per week. score ranges from 0-14; lower scores indicate less achievement of physical activity guidelines
Diet quality | through study completion, 6 months average
  24-hour dietary recall will be collected by study staff, who will use the Automated Self Administered 24 Hour Dietary Recall Assessment Tool (ASA24) to record data for diet quality assessment
Capability | through study completion, 6 months average
  Assessed via the Diabetes Empowerment Scale (DES), a measure of self-efficacy. Average score ranges from 28-140; higher scores indicate greater diabetes empowerment
Healthmine app use | during microrandomized trial, observational period
  Percent of days with app use, per study period will be determined.
Continuous glucose monitor use use | during microrandomized trial, observational period
  Defined as percent of days with CGM data available, per study period.
Motivation to engage in diabetes self-management | through study completion, 6 months average
  Measured via Treatment Self-Regulation Questionnaire (TSRQ). score ranges from 15-105; scoring is based on and average between subscales of intrinsic vs. extrinsic motivation.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | through study completion, 6 months average
  weight and height will be combined to report BMI in kg/m^2
Diabetes distress | through study completion; 6 months average
  Measured via Problem Areas in Diabetes Scale (PAID-5). Score ranges from 0-20; a total score of 8 or more indicates possible diabetes related emotional distress.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen Vajravelu, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, appendices)
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: proposals should be directed to vajravelume@upmc.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years